CLINICAL TRIAL: NCT05111015
Title: Tracking Results of Ablations to Combat AF Registry Generation 2
Acronym: TRAC-AF
Status: Recruiting | Type: Observational
Sponsor: AtriCure, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TRAC-AF Registry
Record Dates: First submitted 2021-10-28; First posted 2021-11-08 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Open Concomitant Surgical Ablation Procedures — AtriCure's Open Concomitant Surgical Ablation Devices used for the management of Atrial Fibrillation.
Device: Hybrid (Convergent) Ablation Procedures — AtriCure's Hybrid (Convergent) Ablation Devices used for the management of Atrial Fibrillation.
Device: AtriCure Hybrid Totally Thoracoscopic Ablation Procedures — AtriCure's Hybrid Totally Thoracoscopic Surgical Ablation Devices used for the management of Atrial Fibrillation.
Device: AtriCure LAA Exclusion Procedures — AtriCure's LAA Exclusion Devices used to exclude the Left Atrial Appendage for the management of Atrial Fibrillation.

SUMMARY:
The primary objective of the TRAC-AF Registry is to capture real-world safety and effectiveness data on AtriCure devices used to conduct open concomitant and/or hybrid ablation, and management of the LAA concomitant to a cardiac ablation.

DETAILED DESCRIPTION:
Up to 10,000 patients at up to 250 sites. Participating regions may include US, Canada, Europe, Asia Pacific and others to be determined. Registry participating sites will enroll patients that meet all inclusion criteria and no exclusion criteria without preselection or bias. Each patient will be followed for a period of up to ten (10) years after their procedure according to the standard practice at the enrolling center. There will be no additional visits, nor procedures, for subjects who participate in the registry.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has been scheduled by physician(s) to undergo or has undergone cardiac ablation procedure(s)
2. Patient is willing to provide informed consent
3. Patient whose age is 18 years or above, or of legal age to give informed consent specific to state and national law

Exclusion Criteria:

1. Other medical, social, or psychological conditions that in the opinion of the Investigator precludes the subject from appropriate consent or adherence to the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The TRAC-AF registry eligibility is open to sites and physicians performing open concomitant or hybrid ablation therapy procedures as treatments for patients diagnosed with paroxysmal, persistent or long-standing persistent atrial fibrillation using at least one of AtriCure's ablation devices. Subjects must have been scheduled to undergo or have undergone the cardiac ablation treatment and must meet all eligibility criteria in order for their treatment and results to be considered for this registry.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2013-02 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Patient's AF burden 6-month after receiving the ablation procedure | 6 months
  Collect patient data on Atrial Fibrillation burden after the ablation procedure as documented by long term event monitoring or identified during the exam after a six-month recovery period.
Adverse events of the ablation procedure as atrial fibrillation management | 1 year
  Collect data on adverse events occurred during and post operation to assess the safety of the ablation procedure.

OTHER OUTCOMES:
Medications | 12 months
  On/Off AAD or Anticoagulant post procedure

CONTACTS AND LOCATIONS:
Locations (28):
- United States (26):
  - Huntsville Hospital, Huntsville, Alabama
  - St. Bernards Medical Center, Jonesboro, Arkansas
  - CHI St. Vincent Heart Institute, Little Rock, Arkansas
  - Loma Linda University Medical Center, Loma Linda, California
  - Adventist Heart Institute (St. Helena Hospital), St. Helena, California
  - Valley View Hospital, Glenwood Springs, Colorado
  - MedStar Washington Hospital, Washington D.C., District of Columbia
  - Delray Medical Center, Delray Beach, Florida
  - University of Florida, Gainesville, Florida
  - Orlando Health Heart & Vascular Institute, Orlando, Florida
  - St. Joseph's Hospital (BayCare), Tampa, Florida
  - Franciscan Health, Indianapolis, Indiana
  - Kansas City Heart Rhythm Institute, Overland Park, Kansas
  - Norton Heart & Vascular Institute, Louisville, Kentucky
  - University of Michigan, Ann Arbor, Michigan
  - Corewell Health, Grand Rapids, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Maimonides Health Heart & Vascular Institute, Brooklyn, New York
  - Vassar Brothers Medical Center, Poughkeepsie, New York
  - Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina
  - UH Cleveland Harrington Heart & Vascular Institute, Cleveland, Ohio
  - Jackson Madison County General Hospital, Jackson, Tennessee
  - Centennial Medical Center, Nashville, Tennessee
  - Michael E. DeBakey VAMC - Houston, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (2):
  - Nova Scotia Health Authority, Halifax, Nova Scotia
  - Waterloo Regional Health Network, Kitchener, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://atricure.com/